CLINICAL TRIAL: NCT06778902
Title: AZA Combined with R-GemOx for the Initial Treatment of Elderly DLBCL: an Open, Single-arm, Multicenter Clinical Study
Brief Title: AZA Combined with R-GemOx for Elderly DLBCL Patients
Acronym: Dragon
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Daping Hospital and the Research Institute of Surgery of the Third Military Medical University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2024-322; ZXYZZKY07 (Other Grant/Funding Number: Army Medical Center Talent Innovation Ability Training Plan)
Record Dates: First submitted 2025-01-07; First posted 2025-01-16 (Actual); Last update posted 2025-01-16 (Actual); Status verified 2024-12

CONDITIONS: DLBCL - Diffuse Large B Cell Lymphoma
Keywords: Diffuse large B-cell lymphoma; GemOx; R; AZA
MeSH Terms: conditions — Dendritic Cell Sarcoma, Interdigitating; Lymphoma, Large B-Cell, Diffuse | interventions — Azacitidine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- AZA+GemOx (Experimental): Elderly DLBCL patients will receive AZA in combination with R-GemOx for a total of 8 treatment cycles (3 weeks per cycle). The efficacy was evaluated every 4 cycles, and if the efficacy was evaluated as complete remission (CR) or partial remission (PR), the original chemotherapy regimen was continued for 4 courses. If efficacy was assessed as stable disease (SD) or progressive disease (PD), the study was withdrawn.After 8 cycles of induction therapy, if the response is assessed as CR or PR, patients may end treatment or receive rituximab maintenance therapy.
  Interventions: Drug: azacytidine; Drug: R-GemOx

INTERVENTIONS:
Drug: azacytidine — Azacytidine: 75mg/m2, d1-d5
Drug: R-GemOx — Rituximab: 375mg/m2, d6; Gemcitabine: 1g/m2, d7 Oxaliplatin: 100mg/m2, d7

SUMMARY:
This is a prospective, single-arm, multicenter, phase II clinical trial to evaluate the efficacy and safety of AZA（azacytidine）combined with the R-GemOx (rituximab, gemcitabine and oxaliplatin) regimen as first-line treatment in elderly diffuse large B-cell lymphoma (DLBCL) patients.

DETAILED DESCRIPTION:
The purpose of this phase II clinical trial is to evaluate the efficacy and safety of AZA in combination with R-GemOx for untreated elderly DLBCL patients.

The induction phase consisted of 8 cycles of AZA in combination with R-GemOx for a total of 8 treatment cycles. The efficacy was evaluated every 4 cycles, and if the efficacy was evaluated as complete remission (CR) or partial remission (PR), the original chemotherapy regimen was continued for 4 courses. If efficacy was assessed as stable disease (SD) or progressive disease (PD), the study was withdrawn.After 8 cycles of induction therapy, if the response is assessed as CR or PR, patients may end treatment or receive rituximab maintenance therapy.

The primary endpoint is the overall response rate (ORR).Secondary efficacy measures included CR and PR,SD, progression-free survival (PFS) and overall survival (OS).

ELIGIBILITY:
Key Inclusion Criteria:

1. Subjects fully understand and voluntarily participate in this study and sign informed consent.
2. Aged ≥60 years, both male and female.
3. Pathologically confirmed DLBCL
4. There must be at least one measurable or evaluable lesion that meets the evaluation criteria for Lugano 2014 lymphoma.
5. No previous chemotherapy or radiotherapy for DLBCL has been received.
6. Expected survival ≥3 months.

Key Exclusion Criteria:

1. DLBCL combined with other types of lymphoma. Transformed DLBCL.
2. DLBCL with central nervous system invasion.
3. The patients have contraindications to any drug in the combined treatment.
4. Patients with the infection of human immunodeficiency virus (HIV) and/or acquired immunodeficiency syndrome.
5. Mentally ill persons or persons unable to obtain informed consent.
6. The investigators think that the patient is not suitable for the study.

Ages: 60 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2025-02-01 (Estimated); Primary Completion 2028-01-01 (Estimated); Study Completion 2028-01-01 (Estimated)

PRIMARY OUTCOMES:
Objective response rate(ORR) | Up to 8 cycles (each cycle is 21 days)
  To investigate the preliminary anti-tumor efficacy

SECONDARY OUTCOMES:
Complete remission(CR) | Up to 8 cycles (each cycle is 21 days)
  To investigate the preliminary anti-tumor efficacy
Partial remission(PR) | Up to 8 cycles (each cycle is 21 days)
  To investigate the preliminary anti-tumor efficacy
Overall Survival (OS) | From the date of enrollment until the date of death from ant cause, assessed up to 24 months
  To investigate the preliminary anti-tumor efficacy
Progression-free survival (PFS) | From the date of enrollment until the date of the first documented progression or date of death from any cause, whichever came first, assessed up to 24 months
  To investigate the preliminary anti-tumor efficacy
Number of participants with adverse events (AE) and severe adverse events (SAE) as assessed by CTCAE v5.0 | Through study completion, an average of 2 years
  To identify the incidence of AE and SAE

OTHER OUTCOMES:
The correlation of gene mutations and alterations in relevant signaling pathways with the efficacy and survival in DLBCL | Through study completion, an average of 2 years
  To explore the correlations between gene mutations and response and prognosis

CONTACTS AND LOCATIONS:
Locations (1):
- Daping Hospital, Third Military Medical University (Army Medical University), Chongqing, China

IPD SHARING:
Plan to Share IPD: No